CLINICAL TRIAL: NCT03235856
Title: Retrospective Digital Computer Analysis of Keratoconus Evolution - REDCAKE
Acronym: REDCAKE
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Principal Investigator, Jos Rozema, Senior researcher, Dpt of Ophthalmology, University Hospital, Antwerp
Other Study IDs: ECR-AS-2017-12
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Keratoconus patients: This study involves a retrospective analysis of data recorded during routine clinical follow-up of keratoconus patients. As such, the impact for the patient is minimal as no additional tests need to be performed

SUMMARY:
The purpose of this study is to create a database of keratoconic eyes with two or more corneal topographies/tomographies, at least 5 months apart

DETAILED DESCRIPTION:
Title: Keratometry values such as K1, K2 and the angle between these two; Value and location of the thinnest corneal point; Pachymetry progression (radial change of pachymetry); IS value (i.e., ratio of average curvature in superior and inferior sections)

Description:

The primary endpoint is to obtain a database, containing at least two valid corneal biometry measurements (Scheimpflug) recorded at least 5 months apart, for a predetermined number of suitable keratoconus patients.

These data will be used to create a personalized three-dimensional model of the cornea at each time point, which permits classifying corneas according to shape and stage, as well as assessing the influence of patient age, gender, family history and ophthalmic habits (e.g. eye rubbing) on keratoconus progression. Based on corneal changes over time, an estimate of the underlying biomechanical changes will be made. All these data will then be combined to develop software for automated keratoconus detection and progression risk assessment to help ophthalmologists decide when to perform crosslinking on their patients.

The primary variables are the elevation parameters derived directly from the Scheimpflug measuring device export files, along with the demographic and medical information (if available).

Time frame: 5 months

Once a predictive model for keratoconus progression speed based on multiple measurements, this can be improved to make predictions based on a single measurement. Furthermore, the database obtained in this work will also be a valuable resource to analyse the variation in keratoconus shape, which may lead to an improved classification of keratoconus types

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-40 years.
* Clinically diagnosed mild or moderate keratoconus in one or both eyes
* Two or more Scheimpflug measurements (type Pentacam HR, Pentacam AXL, Ziemer Galilei, CSO Sirius) of good technical quality, separated at least five months apart.

Exclusion Criteria:

* Corneal scarring present in both eyes.
* Known corneal or retinal pathologies, apart from keratoconus
* Known ocular procedures/ treatments (including crosslinking)
* Known systemic diseases (e.g. diabetes, MS, HIV/AIDS, hypertension,…), except allergies
* Change in contact lenses between measurements (e.g. start wearing lenses, change from corneal to scleral lenses, etc.)
* Fluorescein drops instilled into the eye before Scheimpflug measurement.

Ages: 12 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study involves a retrospective analysis of data recorded during routine clinical follow-up of keratoconus patients. As such, the impact for the patient is minimal as no additions tests need to be performed
Sampling Method: Non-Probability Sample
Enrollment: 972 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
To obtain a database, containing at least two valid corneal Scheimpflug measurements recorded at least 5 months apart, of 1500 keratoconus patients. | 5 months
  These data will be used to create a personalized three-dimensional model of the cornea at each time point, which permits classifying corneas according to shape and stage, as well as assessing the influence of patient age, gender, family history and ophthalmic habits (e.g. eye rubbing) on keratoconus progression. Based on corneal changes over time, an estimate of the underlying biomechanical changes will be made.
To develop software to automatically detect keratoconus and estimate the keratoconus progression speed | 18 months
  The data from Outcome 1 will be combined to develop software for automated keratoconus detection and progression risk assessment to help ophthalmologists decide when to perform cross-linking on their patients.

SECONDARY OUTCOMES:
To improve the predictive model for keratoconus progression speed so it can work using only one single measurement | 18 months
  Once a predictive model for keratoconus progression speed based on multiple measurements, this can be improved to make predictions based on a single measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koppen C, Jimenez-Garcia M, Kreps EO, Ni Dhubhghaill S, Rozema JJ; REDCAKE Study Group. Definitions for Keratoconus Progression and Their Impact on Clinical Practice. Eye Contact Lens. 2024 Jan 1;50(1):1-9. doi: 10.1097/ICL.0000000000001038. Epub 2023 Oct 9. PMID 37816249
- [Derived] Jimenez-Garcia M, Kreps EO, Ni Dhubhghaill S, Koppen C, Rozema JJ; REDCAKE Study Group. Determining the Most Suitable Tomography-Based Parameters to Describe Progression in Keratoconus. The Retrospective Digital Computer Analysis of Keratoconus Evolution Project. Eye Contact Lens. 2021 Sep 1;47(9):486-493. doi: 10.1097/ICL.0000000000000800. PMID 34050086
- [Derived] Jimenez-Garcia M, Ni Dhubhghaill S, Koppen C, Varssano D, Rozema JJ; and The REDCAKE Study Group. Baseline Findings in the Retrospective Digital Computer Analysis of Keratoconus Evolution (REDCAKE) Project. Cornea. 2021 Feb 1;40(2):156-167. doi: 10.1097/ICO.0000000000002389. PMID 32541189